CLINICAL TRIAL: NCT02292771
Title: Randomized, Double-blind, Multicenter, Phase III Study Comparing the Efficacy and Safety of Retosiban Versus Atosiban Therapy for Women in Spontaneous Preterm Labor
Brief Title: A Randomized Study Comparing the Efficacy and Safety of Retosiban Versus Atosiban for Women in Spontaneous Preterm Labour
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was stopped due to the feasibility of recruiting the study in a timely manner
Sponsor: GlaxoSmithKline (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 200721; 2014-001826-13 (EudraCT Number)
Record Dates: First submitted 2014-11-13; First posted 2014-11-17 (Estimated); Results first posted 2018-09-10 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Obstetric Labour, Premature
Keywords: Spontaneous Preterm Labor; retosiban; GSK221149; atosiban
MeSH Terms: conditions — Premature Birth | interventions — GSK221149A; atosiban

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Retosiban + Atosiban Placebo (Experimental): Participants will receive retosiban 6 milligrams (mg) intravenous (IV) loading dose over 5 minutes, followed by a 6mg/hour continuous infusion over 48 hours. For subjects with an inadequate response after the first hour of treatment, investigators will administer another 6mg IV loading dose and increase the infusion rate to 12 mg/hour for the remainder of the 48-hour treatment period. Participants will also receive placebo infusion matched for the atosiban loading (bolus) dose and continuous infusion to ensure blinding.
  Interventions: Drug: Retosiban; Drug: Placebo matching atosiban
- Atosiban + Retosiban Placebo (Active Comparator): Participants will receive atosiban in 3 successive stages: an initial bolus dose (6.75 mg) over 1 minute, immediately followed by a continuous infusion at 18 mg/hour for 3 hours, followed by a 6 mg/hour infusion for the remainder of the 48-hour treatment period. Participants will also receive placebo infusion matched for retosiban loading (bolus) dose and continuous infusion to ensure blinding.
  Interventions: Drug: Atosiban; Drug: Placebo matching retosiban

INTERVENTIONS:
Drug: Retosiban — Solution for infusion, consisting of a clear colorless solution of retosiban at a concentration of 15 milligram/milliliter (mg/mL) in 56% volume/volume ethanol/acetate buffer concentrate supplied in 5 mL vial containing 75mg retosiban.
  Arms: Retosiban + Atosiban Placebo
Drug: Atosiban — Clear, colorless solution for injection in a 0.9-mL vial containing 6.75 mg of atosiban. Clear, colorless concentrate for solution for infusion in a 5-mL vial containing 37.5 mg atosiban.
  Arms: Atosiban + Retosiban Placebo
Drug: Placebo matching retosiban — A placebo infusion containing 0.9% sodium chloride (NaCl) matched for retosiban loading (bolus) dose and continuous infusion.
  Arms: Atosiban + Retosiban Placebo
Drug: Placebo matching atosiban — A placebo infusion containing 0.9% NaCl matched for the atosiban loading (bolus) dose and continuous infusion.
  Arms: Retosiban + Atosiban Placebo

SUMMARY:
The primary objective of this study is to demonstrate the superiority of retosiban to prolong pregnancy in females with spontaneous preterm labor compared with atosiban. This objective is based on the hypothesis that prolonging the time to delivery in the absence of harm may benefit the newborn, particularly in women who experience spontaneous preterm labor at early gestational ages (GA). This study is designed to test this hypothesis through a direct comparison with atosiban, a mixed oxytocin vasopressin antagonist indicated for short-term use to delay imminent preterm birth in women between 24^0/7 and 33^6/7 weeks' gestation in preterm labor. This is a randomized, double-blind, double-dummy study, which consists of 6 phases: Screening, Inpatient Randomized Treatment, Post Infusion Assessment, Delivery, Maternal Post Delivery Assessment, and Neonatal Medical Review. Approximately 330 females will be randomly assigned to retosiban or atosiban treatment in a 1:1 ratio. The duration of any one subject's (maternal or neonatal) participation in the study will be variable and dependent on GA at study entry and the date of delivery.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated written informed consent is required prior to a subject's participation in the study and the performance of any protocol specific procedures. Adolescents aged 12 to 17 years must provide written agreement to participate in the study in accordance with applicable regulatory and country or state requirements. Subjects will also be asked to sign a release for medical records at the time of consenting to allow access to both the maternal and neonatal records including information about delivery and infant care as well as information collected prior to the consent having been signed.
* Females aged 12 to 45 years, with an uncomplicated, singleton pregnancy and intact membranes in preterm labor (Note: This protocol includes pregnant adolescents, aged 12 to 17 years, as appropriate, based on national or local regulations.).
* Gestational age between 24^0/7 and 33^6/7 weeks as determined by known fertilization date, either in vitro fertilization or intrauterine insemination, last menstrual period confirmed by the earliest ultrasound prior to 24^0/7 weeks' gestation, or the earliest ultrasound alone prior to 24^0/7 weeks' gestation, whichever is the most accurate method available for each subject. In situations where prenatal ultrasound records are not available at the time the subject presents, the investigator will make every effort to obtain these records (either via computer records, directly from the subject's primary care obstetrician, or via telephone). However, in cases in which these records are not readily available (e.g., off hours, holiday), it is within the investigator's discretion to use GA based on a verbal history from the subject with the intent of getting confirmation from the medical records as soon as possible.
* Subjects must be diagnosed with preterm labor according to both of the following criteria:

Regular uterine contractions at a rate of >=4 contractions of at least 30 seconds duration during a 30-minute interval confirmed by tocodynamometry

AND at least 1 of the following:

Cervical dilation >=2 centimeter (cm) and <=4 cm by digital cervical examination or If <2 cm dilation by digital cervical examination, a cervical change consisting of an increase of at least 25% effacement or 1 cm dilation

* Treatment naïve subjects and subjects not adequately responding to tocolytics other than atosiban (e.g., transfers from other care units) during their current episode of preterm labor may be eligible for the study. Historical failure of a tocolytic treatment in a previous episode of preterm labor is not a required inclusion criterion. Tocolytic failure is defined by progressive cervical changes or continuing uterine contractions.

Exclusion Criteria:

* Fever with a temperature greater than 100.4°fahrenheit (F) (38°Celcius [C]) for more than 1 hour or >=101°F (38.3°C) in the 24 hours prior to the start of study treatment.
* Women with maternal-fetal conditions that potentially necessitate the need for delivery, such as pre-eclampsia or fetal compromise
* A fetus with any diagnosis, condition, treatment, or other factor that in the opinion of the investigator has the potential to affect or confound assessments of efficacy or safety (e.g., nonreassuring fetal status, intrauterine growth restriction, major congenital anomaly).
* Preterm premature rupture of membranes
* Women with any confirmed or suspected contraindication to prolongation of pregnancy, such as placental abruption, chorioamnionitis, or placenta previa
* Evidence of polyhydramnios (amniotic fluid index [AFI] >25 cm) or oligohydramnios (AFI <5 cm).
* Women with co-morbid medical or obstetric conditions that in the opinion of the investigator have the potential to complicate the pregnancy course and outcomes, such as uncontrolled hypertension, uncontrolled diabetes (if known, history of glycosylated hemoglobin >8% at any time during pregnancy), or compromise the safety of the subject, such as underlying cardiovascular disorder (specifically ischemic cardiac disease, congenital heart disease, pulmonary hypertension, valvular heart disease, arrhythmias, and cardiomyopathy).
* Women with a history of substance abuse or urine drug screen findings suggestive of substance abuse that may either be implicated as the cause of preterm labor (e.g., abuse of cocaine or methamphetamines) or have the potential to complicate the pregnancy outcome (e.g., alcohol abuse or opioid addiction).
* Women with any diagnosis, condition, treatment, or other factor that in the opinion of the investigator has the potential to affect or confound assessments of efficacy or safety.
* Women with documented active hepatitis B or hepatitis C viral infection, unstable liver disease (as defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, or persistent jaundice), cirrhosis, known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of sensitivity to the IPs or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GlaxoSmithKline (GSK)/PPD medical monitor, contraindicates their participation.

Ages: 12 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 97 (Actual)
Dates: Start 2015-03-16 (Actual); Primary Completion 2017-08-25 (Actual); Study Completion 2017-08-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (20):
- Belgium (2):
  - GSK Investigational Site, Bruges
  - GSK Investigational Site, Brussels
- Germany (3):
  - GSK Investigational Site, Freiburg im Breisgau, Baden-Wurttemberg
  - GSK Investigational Site, Jena, Thuringia
  - GSK Investigational Site, Hamburg
- Israel (6):
  - GSK Investigational Site, Haifa
  - GSK Investigational Site, Holon
  - GSK Investigational Site, Kfar Saba
  - GSK Investigational Site, Petah Tikva
  - GSK Investigational Site, Safed
  - GSK Investigational Site, Tel Aviv
- Italy (2):
  - GSK Investigational Site, Siena, Tuscany
  - GSK Investigational Site, Monza
- Mexico (2):
  - GSK Investigational Site, Monterrey, Nuevo León
  - GSK Investigational Site, Ciudad Obregón, Sonora
- South Korea (2):
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Sungnam
- GSK Investigational Site, Zaragoza, Spain
- GSK Investigational Site, Uppsala, Sweden
- GSK Investigational Site, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20389

RESULTS

PARTICIPANT FLOW:
Recruitment Details: ZINN was a randomized, double-blind, double-dummy multicenter study to compare efficacy and safety of retosiban versus atosiban in female participants aged 12 to 45 years with an uncomplicated singleton pregnancy in preterm labor with intact membranes between 24 0/7 and 33 6/7 weeks gestation.
Pre-assignment Details: From 330 planned participants 97 were randomized to receive either retosiban or atosiban intravenous (IV) infusion in a ratio of 1:1. The study was terminated early due to feasibility.
Groups:
- Retosiban: Participants were administered 6 milligram (mg) IV loading dose of retosiban over 5 minutes followed by a 6 milligram per hour (mg/hour) continuous infusion of retosiban over 48 hours. Participants with an inadequate response any time after first hour of treatment were administered another 6 mg retosiban loading dose followed by 12 mg/hour continuous infusion for remainder of 48-hour treatment period.
- Atosiban: Participants were administered atosiban in 3 successive stages. An initial bolus dose of 6.75 mg using atosiban 6.75 mg/0.9 milliliter (mL) solution for injection, followed by continuous high dose infusion at 18 mg/hour for 3 hours, then a lower 6 mg/hour infusion for the remainder of the 48-hour using the atosiban 37.5 mg/5 mL concentrate for solution.
Period: Overall Study
Arm/Group | Retosiban | Atosiban
Started | 47 | 50
Completed | 43 | 48
Not Completed | 4 | 2
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Population: Maternal intent-to-treat (ITT) Population comprised of all mothers randomly assigned to treatment who have been exposed to study treatment irrespective of their compliance to the planned course of treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Retosiban | Atosiban | Total
Number analyzed (Participants) | 47 | 50 | 97
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Maternal intent-to-treat (ITT) Population comprised of all mothers randomly assigned to treatment who have been exposed to study treatment irrespective of their compliance to the planned course of treatment.
  Years | 27.7 (6.15) | 27.1 (5.66) | 27.4 (5.88)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Maternal ITT Population
  Participants
    Female | 47 | 50 | 97
    Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Count of Participants] — Population: Maternal ITT Population
  Count of Participants
    White/Caucasian/European Heritage | 21 | 31 | 52
    American Indian or Alaskan Native | 7 | 4 | 11
    East Asian Heritage | 9 | 4 | 13
    Arabic/North African Heritage | 11 | 10 | 21
    African American/African Heritage | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Time to Delivery From the Start of Investigational Product (IP) Administration
Description: Time to delivery is the number of days from the first dose of study treatment until delivery. The time to delivery was calculated as the days between the delivery and start time of the study treatment infusion using the formula: Time to delivery (days) = (date and time of delivery minus date and time of start of infusion) divided by (24 multiplied by 60). The adjusted mean number of days to delivery along with standard error has been presented. Maternal intent-to-treat (ITT) Population comprised of all mothers randomly assigned to treatment who have been exposed to study treatment irrespective of their compliance to the planned course of treatment.
Time Frame: Up to 17 weeks
Population: Maternal ITT Population
Measure: Mean (Standard Error); unit: Days
Arm/Group | Retosiban | Atosiban
Number analyzed (Participants) | 47 | 50
Days | 32.51 (2.990) | 33.71 (2.531)
Statistical Analysis 1: Comparison: Retosiban vs Atosiban; Test type: Superiority; p = 0.3797, Finite mixture model; Mean Difference (Final Values) = -1.20, 95% CI 2-sided [-8.879 to 6.479]

2. Secondary Outcome: Number of Participants With Births Prior to 37 0/7 Weeks Gestation
Description: Gestational age (GA) at birth (weeks) is defined as the GA when the baby is born. Participants were considered to have delivered prior to 37 0/7 weeks, that is preterm , if the GA at birth is less than 37 0/7 weeks. The number of participants who delivered prior to 37 0/7 weeks gestation has been presented. Logistic regression model was used to calculate p-values.
Time Frame: Up to 13 weeks
Population: Maternal ITT Population
Measure: Number; unit: Participants
Arm/Group | Retosiban | Atosiban
Number analyzed (Participants) | 47 | 50
Participants | 25 | 28
Statistical Analysis 1: Comparison: Retosiban vs Atosiban; Test type: Superiority; p = 0.9520, Regression, Logistic; Odds Ratio (OR) = 1.0, 95% CI 2-sided [0.44 to 2.18]

3. Secondary Outcome: Number of Participants With Births at Term
Description: Participants were considered to have delivered at term if the gestational age was >=37 0/7. The number of participants who delivered at term, that is, 37 0/7 to 41 6/7 weeks gestation has been presented. Logistic regression model was used to calculate p-values.
Time Frame: Up to 17 weeks
Population: Maternal ITT Population
Measure: Number; unit: Participants
Arm/Group | Retosiban | Atosiban
Number analyzed (Participants) | 47 | 50
Participants | 21 | 22
Statistical Analysis 1: Comparison: Retosiban vs Atosiban; Test type: Superiority; p = 0.9520, Regression, Logistic; Odds Ratio (OR) = 1.0, 95% CI 2-sided [0.46 to 2.29]

4. Secondary Outcome: Length of Neonatal Hospital Stay
Description: The length of stay was collected from medical records and was calculated as the days between the delivery date and time and discharge date and time. Log of length of stay was calculated as treatment plus GA at randomization plus established progesterone use based on Analysis of covariance (ANCOVA) model. The p-value was calculated using t-test method. Neonatal ITT Population comprised of all neonates whose mothers were the randomized participants who have been exposed to study treatment, that is, mothers from the ITT Population.
Time Frame: Up to 28 days post estimated date of delivery (EDD) of 40 0/7 weeks gestation
Population: Neonatal ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Days
Arm/Group | Retosiban | Atosiban
Number analyzed (Participants) | 47 | 50
Days | 4.98 [3.54 to 6.99] | 4.38 [3.15 to 6.09]
Statistical Analysis 1: Comparison: Retosiban vs Atosiban; Test type: Superiority; p = 0.5672, ANCOVA; Ratio = 1.14, 95% CI 2-sided [0.73 to 1.76], Standard Error of Mean 0.222

5. Secondary Outcome: Number of Neonates With Composite Neonatal Morbidity and Mortality
Description: The neonatal composite endpoint was determined from review of medical records and included the following components: fetal or neonatal death, Respiratory Distress Syndrome (RDS), bronchopulmonary dysplasia (BPD), necrotizing enterocolitis (NEC) or isolated perforation, sepsis based on positive blood culture with clinical features of sepsis, meningitis based on positive results for cerebrospinal fluid culture performed as part of infection workup, retinopathy of prematurity (ROP), Intraventricular Hemorrhage (IVH), white matter injury and cerebellar hemorrhage.
Time Frame: Up to 28 weeks after EDD (40 weeks gestation)
Population: Neonatal ITT Population
Measure: Number; unit: Participants
Arm/Group | Retosiban | Atosiban
Number analyzed (Participants) | 47 | 50
Participants | 3 | 2
Statistical Analysis 1: Comparison: Retosiban vs Atosiban; Test type: Superiority; p = 0.5066, Regression, Logistic; Odds Ratio (OR) = 1.9, 95% CI 2-sided [0.30 to 11.71]

6. Secondary Outcome: Number of Neonates With Any Composite Neonatal Morbidity and Mortality, Excluding RDS
Description: The neonatal composite endpoint was determined from review of medical records and included the following components: fetal or neonatal death, RDS, BPD, NEC or isolated perforation, sepsis based on positive blood culture with clinical features of sepsis, meningitis based on positive results for cerebrospinal fluid culture performed as part of infection workup, ROP, IVH, white matter injury and cerebellar hemorrhage. Number of neonates with any composite neonatal morbidity and mortality component, excluding RDS has been presented.
Time Frame: Up to 28 weeks after EDD (40 weeks gestation)
Population: Neonatal ITT Population
Measure: Number; unit: Participants
Arm/Group | Retosiban | Atosiban
Number analyzed (Participants) | 47 | 50
Participants | 0 | 1

7. Secondary Outcome: Number of Neonates With Each Individual Component of Composite Neonatal Morbidity and Mortality
Description: The neonatal composite endpoint was determined from review of medical records and included the following components: fetal or neonatal death, RDS, BPD, NEC or isolated perforation, sepsis based on positive blood culture with clinical features of sepsis, meningitis based on positive results for cerebrospinal fluid culture performed as part of infection workup, ROP, IVH, cerebellar hemorrhage and white matter injury included Periventricular Leukomalacia PVL), porencephalic cyst, and persistent ventriculomegaly. Number of neonates with with each individual component of the composite neonatal morbidity and mortality has been presented.
Time Frame: Up to 28 weeks after EDD (40 weeks gestation)
Population: Neonatal ITT Population
Measure: Number; unit: Participants
Arm/Group | Retosiban | Atosiban
Number analyzed (Participants) | 47 | 50
Participants
  Fetal death | 0 | 0
  Neonatal death | 0 | 1
  RDS | 3 | 1
  BPD | 0 | 0
  NEC or isolated perforation | 0 | 0
  Sepsis | 0 | 0
  Meningitis | 0 | 0
  ROP | 0 | 0
  IVH | 0 | 0
  PVL | 0 | 0
  Porencephalic Cyst | 0 | 0
  Persistent Ventriculomegaly | 0 | 0
  Cerebellar Hemorrhage | 0 | 0

8. Secondary Outcome: Length of Stay in Specialized Care Unit
Description: Length of neonatal stay in specialized care unit like Intensive Care Unit (ICU) or Neonatal Intensive Care Unit (NICU) are reported.
Time Frame: Up to 28 days post EDD (40 0/7 weeks gestation)
Population: Neonatal Safety Population
Measure: Median (Full Range); unit: Days
Arm/Group | Retosiban | Atosiban
Number analyzed (Participants) | 47 | 50
Days | 13.65 [3.5 to 57.5] | 12.49 [7.6 to 21.8]

9. Secondary Outcome: Number of Newborn Participants With Hospital Readmission
Description: Newborn hospital readmission following hospitalization for birth was obtained from the newborn's medical records. Only those participants with data available at the specified data points were analyzed.
Time Frame: Up to 28 days of EDD (40 0/7 weeks gestation)
Population: Neonatal Safety Population
Measure: Number; unit: Participants
Arm/Group | Retosiban | Atosiban
Number analyzed (Participants) | 46 | 50
Participants | 2 | 3

10. Secondary Outcome: Number of Participants With Births Prior to 28 0/7 Weeks Gestation
Description: The number of participants who delivered prior to 28 0/7 weeks gestation has been presented. Only those maternal participants who were randomized prior to 28 0/7 week's gestation and delivered were included.
Time Frame: Up to 4 weeks
Population: Maternal ITT Population
Measure: Number; unit: Participants
Arm/Group | Retosiban | Atosiban
Number analyzed (Participants) | 47 | 50
Participants | 0 | 0

11. Secondary Outcome: Number of Participants With Births Prior to 32 0/7 Weeks Gestation
Description: Number of participants who delivered prior to 32 0/7 weeks gestation has been presented. Only those maternal participants who were randomized prior to 32 0/7 week's gestation and delivered were included.
Time Frame: Up to 8 weeks
Population: Maternal ITT Population
Measure: Number; unit: Participants
Arm/Group | Retosiban | Atosiban
Number analyzed (Participants) | 47 | 50
Participants | 3 | 3
Statistical Analysis 1: Comparison: Retosiban vs Atosiban; Test type: Superiority; p = 0.7790, Regression, Logistic; Odds Ratio (OR) = 0.8, 95% CI 2-sided [0.12 to 4.84]

12. Secondary Outcome: Number of Participants With Births Prior to 35 0/7 Weeks Gestation
Description: Number of participants who delivered prior to 35 0/7 weeks gestation has been presented. Only those maternal participants who were randomized prior to 35 0/7 week's gestation and delivered were included.
Time Frame: Up to 11 weeks
Population: Maternal ITT Population
Measure: Number; unit: Participants
Arm/Group | Retosiban | Atosiban
Number analyzed (Participants) | 47 | 50
Participants | 14 | 14
Statistical Analysis 1: Comparison: Retosiban vs Atosiban; Test type: Superiority; p = 0.6646, Regression, Logistic; Odds Ratio (OR) = 1.2, 95% CI 2-sided [0.51 to 2.90]

13. Secondary Outcome: Number of Participants With Births <=7 Days From the First Study Treatment
Description: Number of participants who delivered in less than or equal to 7 days from first dose of study treatment has been presented.
Time Frame: Up to 7 days
Population: Maternal ITT Population
Measure: Number; unit: Participants
Arm/Group | Retosiban | Atosiban
Number analyzed (Participants) | 47 | 50
Participants | 10 | 7
Statistical Analysis 1: Comparison: Retosiban vs Atosiban; Test type: Superiority; p = 0.1432, Regression, Logistic; Odds Ratio (OR) = 2.3, 95% CI 2-sided [0.75 to 7.24]

14. Secondary Outcome: Number of Participants With Births <=48 Hours From the First Study Treatment
Description: Number of participants who delivered in less than or equal to 48 hours from first dose of study treatment has been presented.
Time Frame: Up to 48 hours
Population: Maternal ITT Population
Measure: Number; unit: Participants
Arm/Group | Retosiban | Atosiban
Number analyzed (Participants) | 47 | 50
Participants | 6 | 6
Statistical Analysis 1: Comparison: Retosiban vs Atosiban; Test type: Superiority; p = 0.5250, Regression, Logistic; Odds Ratio (OR) = 1.5, 95% CI 2-sided [0.43 to 5.15]

15. Secondary Outcome: Number of Participants With Births <=24 Hours From the First Study Treatment
Description: Number of participants who delivered in less than or equal to 24 hours from first dose of study treatment has been presented.
Time Frame: Up to 24 hours
Population: Maternal ITT Population
Measure: Number; unit: Participants
Arm/Group | Retosiban | Atosiban
Number analyzed (Participants) | 47 | 50
Participants | 3 | 6
Statistical Analysis 1: Comparison: Retosiban vs Atosiban; Test type: Superiority; p = 0.4682, Regression, Logistic; Odds Ratio (OR) = 0.6, 95% CI 2-sided [0.13 to 2.58]

16. Secondary Outcome: Number of Maternal Participants With Non-serious Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose: results in death; is life threatening; requires hospitalization or prolongation of existing hospitalization; results in disability/incapacity; is a congenital anomaly/birth defect; important medical events that may require medical or surgical intervention to prevent one of the other outcomes described before; is associated with liver injury and impaired liver function. Maternal Safety Population comprised of all mothers randomly assigned to treatment who have been exposed to study treatment. The number of maternal participants who experienced at least one non-serious AE and one SAE has been presented.
Time Frame: Up to 6 weeks after delivery
Population: Maternal Safety Population
Measure: Number; unit: Participants
Arm/Group | Retosiban | Atosiban
Number analyzed (Participants) | 47 | 50
Participants
  Non-serious AE | 34 | 25
  SAE | 7 | 9

17. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure (DBP) and Systolic Blood Pressure (SBP) in Maternal Participants
Description: SBP and DBP were measured during inpatient randomized treatment phase (15 to 30 minutes, 4 to 8 hours, and 20 to 24 hours after the start of the infusion, at the end of the infusion) and at the post-infusion assessment. Baseline is the last available assessment prior to first dose of study treatment. Change from Baseline is the post-dose visit value minus Baseline. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title).
Time Frame: Baseline and up to 1 week
Population: Maternal Safety Population
Measure: Mean (Standard Deviation); unit: Millimeter of mercury (mmHg)
Arm/Group | Retosiban | Atosiban
Number analyzed (Participants) | 47 | 50
Millimeter of mercury (mmHg)
  DBP; Day 1: 15 to 30 minutes, n=42,45: number analyzed (Participants) | 42 | 45
  DBP; Day 1: 15 to 30 minutes, n=42,45 | -3.6 (10.96) | -0.7 (8.95)
  DBP; Day 1: 4 to 8 hours, n=42,43: number analyzed (Participants) | 42 | 43
  DBP; Day 1: 4 to 8 hours, n=42,43 | -4.3 (11.07) | -3.7 (10.28)
  DBP; Day 1: 20 to 24 hours, n=38,41: number analyzed (Participants) | 38 | 41
  DBP; Day 1: 20 to 24 hours, n=38,41 | -5.7 (9.31) | -4.1 (9.90)
  DBP; Day 2, n=40,42: number analyzed (Participants) | 40 | 42
  DBP; Day 2, n=40,42 | -4.4 (9.57) | -2.6 (9.93)
  DBP; Post-infusion assessment, n=35,41: number analyzed (Participants) | 35 | 41
  DBP; Post-infusion assessment, n=35,41 | -1.6 (8.63) | 1.3 (10.12)
  SBP; Day 1: 15 to 30 minutes, n=42,45: number analyzed (Participants) | 42 | 45
  SBP; Day 1: 15 to 30 minutes, n=42,45 | -2.5 (9.53) | -0.4 (11.02)
  SBP; Day 1: 4 to 8 hours, n=42,43: number analyzed (Participants) | 42 | 43
  SBP; Day 1: 4 to 8 hours, n=42,43 | -4.3 (9.05) | -3.3 (12.21)
  SBP; Day 1: 20 to 24 hours, n=38,41: number analyzed (Participants) | 38 | 41
  SBP; Day 1: 20 to 24 hours, n=38,41 | -4.1 (10.16) | -5.2 (13.03)
  SBP; Day 2, n=40,42: number analyzed (Participants) | 40 | 42
  SBP; Day 2, n=40,42 | -3.9 (11.53) | -3.0 (11.35)
  SBP; Post-infusion assessment, n=35,41: number analyzed (Participants) | 35 | 41
  SBP; Post-infusion assessment, n=35,41 | -1.5 (11.04) | -2.1 (11.37)

18. Secondary Outcome: Change From Baseline in Heart Rate in Maternal Participants
Description: Heart rate was measured during inpatient randomized treatment phase (15 to 30 minutes, 4 to 8 hours, and 20 to 24 hours after the start of the infusion, at the end of the infusion) and at the post-infusion assessment. Baseline is the last available assessment prior to first dose of study treatment. Change from Baseline is the post-dose visit value minus Baseline. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title).
Time Frame: Baseline and up to 1 week
Population: Maternal Safety Population
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Retosiban | Atosiban
Number analyzed (Participants) | 47 | 50
Beats per minute
  Day 1: 15 to 30 minutes, n=42,46: number analyzed (Participants) | 42 | 46
  Day 1: 15 to 30 minutes, n=42,46 | -3.0 (12.65) | -0.8 (10.45)
  Day 1: 4 to 8 hours, n=42, 43: number analyzed (Participants) | 42 | 43
  Day 1: 4 to 8 hours, n=42, 43 | -5.0 (13.69) | -3.0 (13.65)
  Day 1: 20 to 24 hours, n=38, 41: number analyzed (Participants) | 38 | 41
  Day 1: 20 to 24 hours, n=38, 41 | -1.2 (14.44) | -3.1 (13.82)
  Day 2, n=39, 41: number analyzed (Participants) | 39 | 41
  Day 2, n=39, 41 | -2.2 (11.81) | -2.3 (13.44)
  Post-infusion assessment, n=35, 41: number analyzed (Participants) | 35 | 41
  Post-infusion assessment, n=35, 41 | -2.7 (12.90) | -1.8 (13.83)

19. Secondary Outcome: Change From Baseline in Respiratory Rate in Maternal Participants
Description: Respiratory rate was measured during inpatient randomized treatment phase (15 to 30 minutes, 4 to 8 hours, and 20 to 24 hours after the start of the infusion, at the end of the infusion) and at the post-infusion assessment. Baseline is the last available assessment prior to first dose of study treatment. Change from Baseline is the post-dose visit value minus Baseline. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title).
Time Frame: Baseline and up to 1 week
Population: Maternal Safety Population
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Retosiban | Atosiban
Number analyzed (Participants) | 47 | 50
breaths per minute
  Day 1: 15 to 30 minutes, n=25, 28: number analyzed (Participants) | 25 | 28
  Day 1: 15 to 30 minutes, n=25, 28 | 0.3 (2.82) | -0.6 (1.93)
  Day 1: 4 to 8 hours, n=23, 24: number analyzed (Participants) | 23 | 24
  Day 1: 4 to 8 hours, n=23, 24 | 0.0 (1.65) | -0.8 (2.33)
  Day 1: 20 to 24 hours, n=21, 21: number analyzed (Participants) | 21 | 21
  Day 1: 20 to 24 hours, n=21, 21 | 0.2 (1.87) | -0.6 (2.40)
  Day 2, n=23, 24: number analyzed (Participants) | 23 | 24
  Day 2, n=23, 24 | -0.3 (1.64) | 0.2 (3.45)
  Post-infusion assessment, n=22, 23: number analyzed (Participants) | 22 | 23
  Post-infusion assessment, n=22, 23 | -0.3 (2.15) | -1.3 (2.70)

20. Secondary Outcome: Change From Baseline in Temperature in Maternal Participants
Description: Temperature was measured during inpatient randomized treatment phase (15 to 30 minutes, 4 to 8 hours, and 20 to 24 hours after the start of the infusion, at the end of the infusion) and at the post-infusion assessment. Baseline is the last available assessment prior to first dose of study treatment. Change from Baseline is the post-dose visit value minus Baseline. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title).
Time Frame: Baseline and up to 1 week
Population: Maternal Safety Population
Measure: Mean (Standard Deviation); unit: degree Celsius
Arm/Group | Retosiban | Atosiban
Number analyzed (Participants) | 47 | 50
degree Celsius
  Day 1: 15 to 30 minutes, n=41, 43: number analyzed (Participants) | 41 | 43
  Day 1: 15 to 30 minutes, n=41, 43 | -0.02 (0.379) | 0.02 (0.467)
  Day 1: 4 to 8 hours, n=40, 42: number analyzed (Participants) | 40 | 42
  Day 1: 4 to 8 hours, n=40, 42 | -0.06 (0.359) | 0.00 (0.507)
  Day 1: 20 to 24 hours, n=37, 41: number analyzed (Participants) | 37 | 41
  Day 1: 20 to 24 hours, n=37, 41 | -0.07 (0.366) | -0.03 (0.486)
  Day 2, n=40, 42: number analyzed (Participants) | 40 | 42
  Day 2, n=40, 42 | -0.07 (0.467) | -0.06 (0.353)
  Post-infusion assessment, n=35, 41: number analyzed (Participants) | 35 | 41
  Post-infusion assessment, n=35, 41 | -0.18 (0.334) | -0.20 (0.422)

21. Secondary Outcome: Change From Baseline in Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils, Platelets and Leukocytes Count in Maternal Participants
Description: Blood samples were collected for the evaluation of change in basophils, eosinophils, lymphocytes, monocytes, neutrophils, platelets and leukocytes count. Baseline is defined as the last available assessment prior to the first dose of study treatment. Change from Baseline is the post-dose visit value minus Baseline. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title). NA indicates standard deviation was not calculable for a single data point.
Time Frame: Baseline and up to 1 week
Population: Maternal Safety Population
Measure: Mean (Standard Deviation); unit: Billion cells per liter (L)
Arm/Group | Retosiban | Atosiban
Number analyzed (Participants) | 47 | 50
Billion cells per liter (L)
  Basophils;Day2,n=21,23: number analyzed (Participants) | 21 | 23
  Basophils;Day2,n=21,23 | 0.003 (0.0362) | 0.010 (0.0304)
  Basophils;Post-infusion assessment,n=24,28: number analyzed (Participants) | 24 | 28
  Basophils;Post-infusion assessment,n=24,28 | 0.001 (0.0315) | 0.007 (0.0181)
  Basophils;early withdrawal,n=1,1: number analyzed (Participants) | 1 | 1
  Basophils;early withdrawal,n=1,1 | -0.020 (NA) — NA indicates standard deviation was not calculable for a single data point. | 0.030 (NA) — NA indicates standard deviation was not calculable for a single data point.
  Eosinophils;Day2,n=21,23: number analyzed (Participants) | 21 | 23
  Eosinophils;Day2,n=21,23 | -0.010 (0.0626) | -0.037 (0.1181)
  Eosinophils;Post-infusion assessment,n=24,28: number analyzed (Participants) | 24 | 28
  Eosinophils;Post-infusion assessment,n=24,28 | 0.023 (0.0442) | 0.066 (0.1535)
  Eosinophils;early withdrawal,n=1,1: number analyzed (Participants) | 1 | 1
  Eosinophils;early withdrawal,n=1,1 | 0.030 (NA) — NA indicates standard deviation was not calculable for a single data point. | 0.050 (NA) — NA indicates standard deviation was not calculable for a single data point.
  Lymphocytes;Day2,n=21,23: number analyzed (Participants) | 21 | 23
  Lymphocytes;Day2,n=21,23 | 0.186 (0.9115) | 0.067 (0.6017)
  Lymphocytes;Post-infusion assessment,n=24,28: number analyzed (Participants) | 24 | 28
  Lymphocytes;Post-infusion assessment,n=24,28 | 0.348 (0.8611) | 0.233 (0.8047)
  Lymphocytes;early withdrawal,n=1,1: number analyzed (Participants) | 1 | 1
  Lymphocytes;early withdrawal,n=1,1 | 0.270 (NA) — NA indicates standard deviation was not calculable for a single data point. | -1.770 (NA) — NA indicates standard deviation was not calculable for a single data point.
  Monocytes;Day2,n=21,23: number analyzed (Participants) | 21 | 23
  Monocytes;Day2,n=21,23 | 0.082 (0.2222) | 0.044 (0.2702)
  Monocytes;Post-infusion assessment,n=24,28: number analyzed (Participants) | 24 | 28
  Monocytes;Post-infusion assessment,n=24,28 | 0.222 (0.1904) | 0.133 (0.3467)
  Monocytes;early withdrawal,n=1,1: number analyzed (Participants) | 1 | 1
  Monocytes;early withdrawal,n=1,1 | -0.160 (NA) — NA indicates standard deviation was not calculable for a single data point. | 0.410 (NA) — NA indicates standard deviation was not calculable for a single data point.
  Neutrophils;Day2,n=21,23: number analyzed (Participants) | 21 | 23
  Neutrophils;Day2,n=21,23 | 0.102 (2.6712) | 0.559 (3.3890)
  Neutrophils;Post-infusion assessment,n=24,28: number analyzed (Participants) | 24 | 28
  Neutrophils;Post-infusion assessment,n=24,28 | -1.865 (2.9246) | -0.670 (2.7063)
  Neutrophils;early withdrawal,n=1,1: number analyzed (Participants) | 1 | 1
  Neutrophils;early withdrawal,n=1,1 | -0.710 (NA) — NA indicates standard deviation was not calculable for a single data point. | -3.550 (NA) — NA indicates standard deviation was not calculable for a single data point.
  Platelets;Day2,n=22,25: number analyzed (Participants) | 22 | 25
  Platelets;Day2,n=22,25 | 0.0 (25.95) | -2.4 (36.59)
  Platelets;Post-infusion assessment,n=24,31: number analyzed (Participants) | 24 | 31
  Platelets;Post-infusion assessment,n=24,31 | 21.5 (63.14) | 20.6 (43.74)
  Platelets;early withdrawal,n=1,1: number analyzed (Participants) | 1 | 1
  Platelets;early withdrawal,n=1,1 | -33.0 (NA) — NA indicates standard deviation was not calculable for a single data point. | -58.0 (NA) — NA indicates standard deviation was not calculable for a single data point.
  Leukocytes;Day2,n=23,25: number analyzed (Participants) | 23 | 25
  Leukocytes;Day2,n=23,25 | 0.17 (2.785) | 0.72 (2.905)
  Leukocytes;Post-infusion assessment,n=25,30: number analyzed (Participants) | 25 | 30
  Leukocytes;Post-infusion assessment,n=25,30 | -1.18 (2.492) | -0.05 (2.756)
  Leukocytes;early withdrawal,n=1,1: number analyzed (Participants) | 1 | 1
  Leukocytes;early withdrawal,n=1,1 | -0.60 (NA) — NA indicates standard deviation was not calculable for a single data point. | -4.80 (NA) — NA indicates standard deviation was not calculable for a single data point.

22. Secondary Outcome: Change From Baseline in Erythrocytes in Maternal Participants
Description: Blood samples were collected for the evaluation of change in erythrocytes from Baseline. Baseline is defined as the last available assessment prior to the first dose of study treatment. Change from Baseline is the post-dose visit value minus Baseline. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title). NA indicates standard deviation was not calculable for a single data point.
Time Frame: Baseline and up to 1 week
Population: Maternal Safety Population
Measure: Mean (Standard Deviation); unit: Trillion cells per liter
Arm/Group | Retosiban | Atosiban
Number analyzed (Participants) | 47 | 50
Trillion cells per liter
  Day 2, n=23, 27: number analyzed (Participants) | 23 | 27
  Day 2, n=23, 27 | -0.22 (0.284) | -0.29 (0.261)
  Post-infusion assessment, n=25, 31: number analyzed (Participants) | 25 | 31
  Post-infusion assessment, n=25, 31 | 0.06 (0.257) | 0.05 (0.236)
  Early withdrawal, n =1, 1: number analyzed (Participants) | 1 | 1
  Early withdrawal, n =1, 1 | -0.20 (NA) — NA indicates standard deviation was not calculable for a single data point. | -0.70 (NA) — NA indicates standard deviation was not calculable for a single data point.

23. Secondary Outcome: Change From Baseline in Hemoglobin and Erythrocyte Mean Corpuscular Hemoglobin Concentration (MCHC) in Maternal Participants
Description: Blood samples were collected for the evaluation of change in hemoglobin levels and MCHC from Baseline. Baseline is defined as the last available assessment prior to the first dose of study treatment. Change from Baseline is the post-dose visit value minus. NA indicates standard deviation was not calculable for a single data point.
Time Frame: Baseline and up to 1 week
Population: Maternal Safety Population
Measure: Mean (Standard Deviation); unit: grams per liter (g/L)
Arm/Group | Retosiban | Atosiban
Number analyzed (Participants) | 47 | 50
grams per liter (g/L)
  Hemoglobin; Day2, n=23, 27: number analyzed (Participants) | 23 | 27
  Hemoglobin; Day2, n=23, 27 | -5.4 (7.81) | -8.4 (6.86)
  Hemoglobin; Post-infusion assessment, n=25, 31: number analyzed (Participants) | 25 | 31
  Hemoglobin; Post-infusion assessment, n=25, 31 | 0.8 (7.55) | 0.5 (5.37)
  Hemoglobin; early withdrawal, n=1, 1: number analyzed (Participants) | 1 | 1
  Hemoglobin; early withdrawal, n=1, 1 | -8.0 (NA) — NA indicates standard deviation was not calculable for a single data point. | -19.0 (NA) — NA indicates standard deviation was not calculable for a single data point.
  MCHC; Day 2, n=23, 27: number analyzed (Participants) | 23 | 27
  MCHC; Day 2, n=23, 27 | 1.0 (9.41) | 0.9 (6.85)
  MCHC; Post-infusion assessment, n=25, 31: number analyzed (Participants) | 25 | 31
  MCHC; Post-infusion assessment, n=25, 31 | 1.0 (7.36) | 0.4 (8.98)
  MCHC; early withdrawal, n=1, 1: number analyzed (Participants) | 1 | 1
  MCHC; early withdrawal, n=1, 1 | -3.0 (NA) — NA indicates standard deviation was not calculable for a single data point. | 24.0 (NA) — NA indicates standard deviation was not calculable for a single data point.

24. Secondary Outcome: Change From Baseline in Erythrocyte Mean Corpuscular Volume (MCV) and Mean Platelet Volume (MPV) in Maternal Participants
Description: Blood samples were collected for the evaluation of change in MCV and MPV from Baseline. Baseline is defined as the last available assessment prior to the first dose of study treatment. Change from Baseline is the post-dose visit value minus Baseline. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title). NA indicates standard deviation was not calculable for a single data point.
Time Frame: Baseline and up to 1 week
Population: Maternal Safety Population
Measure: Mean (Standard Deviation); unit: femtoliter (fL)
Arm/Group | Retosiban | Atosiban
Number analyzed (Participants) | 47 | 50
femtoliter (fL)
  MCV; Day 2, n=23, 27: number analyzed (Participants) | 23 | 27
  MCV; Day 2, n=23, 27 | 0.3 (2.67) | -0.4 (1.82)
  MCV; Post-infusion assessment, n=25, 31: number analyzed (Participants) | 25 | 31
  MCV; Post-infusion assessment, n=25, 31 | -1.2 (2.17) | -1.0 (2.22)
  MCV; early withdrawal, n=1, 1: number analyzed (Participants) | 1 | 1
  MCV; early withdrawal, n=1, 1 | -1.0 (NA) — NA indicates standard deviation was not calculable for a single data point. | -5.0 (NA) — NA indicates standard deviation was not calculable for a single data point.
  MPV; Day 2, n=22, 25: number analyzed (Participants) | 22 | 25
  MPV; Day 2, n=22, 25 | 0.05 (0.607) | 0.06 (0.553)
  MPV, Post-infusion assessment, n=24, 31: number analyzed (Participants) | 24 | 31
  MPV, Post-infusion assessment, n=24, 31 | -0.10 (0.639) | -0.03 (0.803)
  MPV, early withdrawal, n=1, 1: number analyzed (Participants) | 1 | 1
  MPV, early withdrawal, n=1, 1 | 0.00 (NA) — NA indicates standard deviation was not calculable for a single data point. | -1.40 (NA) — NA indicates standard deviation was not calculable for a single data point.

25. Secondary Outcome: Change From Baseline in Alkaline Phosphatase (ALP), Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), Gamma Glutamyl Transferase (GGT) and Lactate Dehydrogenase (LDH) Levels in Maternal Participants
Description: Blood samples were collected for the evaluation of change in ALP, ALT, AST, GGT and LDH from Baseline. Baseline is defined as the last available assessment prior to the first dose of study treatment. Change from Baseline is the post-dose visit value minus Baseline. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title). NA indicates standard deviation was not calculable for a single data point.
Time Frame: Baseline and up to 1 week
Population: Maternal Safety Population
Measure: Mean (Standard Deviation); unit: International Units per liter (IU/L)
Arm/Group | Retosiban | Atosiban
Number analyzed (Participants) | 47 | 50
International Units per liter (IU/L)
  ALP; Day 2, n=35, 35: number analyzed (Participants) | 35 | 35
  ALP; Day 2, n=35, 35 | -10.1 (12.12) | -12.6 (13.07)
  ALP; Post-infusion assessment, n=30, 35: number analyzed (Participants) | 30 | 35
  ALP; Post-infusion assessment, n=30, 35 | 14.1 (39.85) | 5.9 (15.87)
  ALP; early withdrawal, n=1, 1: number analyzed (Participants) | 1 | 1
  ALP; early withdrawal, n=1, 1 | -6.0 (NA) — NA indicates standard deviation was not calculable for a single data point. | -19.0 (NA) — NA indicates standard deviation was not calculable for a single data point.
  AST; Day 2, n=34, 35: number analyzed (Participants) | 34 | 35
  AST; Day 2, n=34, 35 | -0.9 (4.82) | -1.7 (3.07)
  AST; Post-infusion assessmet, n=29, 35: number analyzed (Participants) | 29 | 35
  AST; Post-infusion assessmet, n=29, 35 | -1.3 (4.87) | -1.3 (4.09)
  AST; early withdrawal, n=1, 1: number analyzed (Participants) | 1 | 1
  AST; early withdrawal, n=1, 1 | -3.0 (NA) — NA indicates standard deviation was not calculable for a single data point. | 1.0 (NA) — NA indicates standard deviation was not calculable for a single data point.
  ALT; Day 2, n= 35, 35: number analyzed (Participants) | 35 | 35
  ALT; Day 2, n= 35, 35 | -0.2 (2.53) | 0.0 (2.40)
  ALT; Post-infusion assessment, n= 30, 35: number analyzed (Participants) | 30 | 35
  ALT; Post-infusion assessment, n= 30, 35 | 0.0 (6.34) | 0.8 (6.19)
  ALT; early withdrawal, n= 1, 1: number analyzed (Participants) | 1 | 1
  ALT; early withdrawal, n= 1, 1 | -2.0 (NA) — NA indicates standard deviation was not calculable for a single data point. | 5.0 (NA) — NA indicates standard deviation was not calculable for a single data point.
  GGT; Day 2, n= 35, 35: number analyzed (Participants) | 35 | 35
  GGT; Day 2, n= 35, 35 | -0.4 (2.44) | -0.9 (3.08)
  GGT; Post-infusion assessment, n=30, 35: number analyzed (Participants) | 30 | 35
  GGT; Post-infusion assessment, n=30, 35 | 17.6 (79.05) | 2.3 (4.39)
  GGT; eearly withdrawal, n=1, 1: number analyzed (Participants) | 1 | 1
  GGT; eearly withdrawal, n=1, 1 | 0.0 (NA) — NA indicates standard deviation was not calculable for a single data point. | 0.0 (NA) — NA indicates standard deviation was not calculable for a single data point.
  LDH; Day 2, n=34, 35: number analyzed (Participants) | 34 | 35
  LDH; Day 2, n=34, 35 | -9.7 (50.58) | -20.0 (29.18)
  LDH; Post-infusion assessment, n=29, 35: number analyzed (Participants) | 29 | 35
  LDH; Post-infusion assessment, n=29, 35 | -2.4 (22.08) | -5.4 (30.93)
  LDH; early withdrawal, n=1, 1: number analyzed (Participants) | 1 | 1
  LDH; early withdrawal, n=1, 1 | -18.0 (NA) — NA indicates standard deviation was not calculable for a single data point. | -59.0 (NA) — NA indicates standard deviation was not calculable for a single data point.

26. Secondary Outcome: Change From Baseline in Albumin and Protein Levels in Maternal Participants
Description: Blood samples were collected for the evaluation of change in albumin and protein levels from Baseline. Baseline is defined as the last available assessment prior to the first dose of study treatment. Change from Baseline is the post-dose visit value minus Baseline. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title). NA indicates standard deviation was not calculable for a single data point.
Time Frame: Baseline and up to 1 week
Population: Maternal Safety Population
Measure: Mean (Standard Deviation); unit: grams per liter (g/L)
Arm/Group | Retosiban | Atosiban
Number analyzed (Participants) | 47 | 50
grams per liter (g/L)
  Albumin; Day 2, n=35, 35: number analyzed (Participants) | 35 | 35
  Albumin; Day 2, n=35, 35 | -1.9 (2.28) | -2.0 (1.95)
  Albumin; Post-infusion assessment, n=30, 35: number analyzed (Participants) | 30 | 35
  Albumin; Post-infusion assessment, n=30, 35 | 0.3 (2.39) | -0.2 (2.26)
  Albumin; early withdrawal, n=1, 1: number analyzed (Participants) | 1 | 1
  Albumin; early withdrawal, n=1, 1 | -4.0 (NA) — NA indicates standard deviation was not calculable for a single data point. | -8.0 (NA) — NA indicates standard deviation was not calculable for a single data point.
  Protein; Day 2, n=35, 35: number analyzed (Participants) | 35 | 35
  Protein; Day 2, n=35, 35 | -3.7 (4.18) | -3.3 (3.69)
  Protein; Post-infusion assessment, n=30, 35: number analyzed (Participants) | 30 | 35
  Protein; Post-infusion assessment, n=30, 35 | 0.5 (4.73) | 0.0 (4.05)
  Protein; early withdrawal, n=1, 1: number analyzed (Participants) | 1 | 1
  Protein; early withdrawal, n=1, 1 | -5.0 (NA) — NA indicates standard deviation was not calculable for a single data point. | -12.0 (NA) — NA indicates standard deviation was not calculable for a single data point.

27. Secondary Outcome: Change From Baseline in Calcium, Chloride, Carbon Dioxide, Glucose, Potassium, Magnesium, Phosphate and Sodium Level in Maternal Participants
Description: Blood samples were collected for the evaluation of change from Baseline in levels of calcium, chloride, carbon dioxide, glucose, potassium, magnesium, phosphate, and sodium. Baseline is defined as the last available assessment prior to the first dose of study treatment. Change from Baseline is the post-dose visit value minus Baseline. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title). NA indicates standard deviation was not calculable for a single data point.
Time Frame: Baseline and up to 1 week
Population: Maternal Safety Population
Measure: Mean (Standard Deviation); unit: millimoles per liter (mmol/L)
Arm/Group | Retosiban | Atosiban
Number analyzed (Participants) | 47 | 50
millimoles per liter (mmol/L)
  Calcium; Day 2, n=34, 35: number analyzed (Participants) | 34 | 35
  Calcium; Day 2, n=34, 35 | -0.097 (0.1125) | -0.078 (0.0884)
  Calcium; Post-infusion assessment, n=29, 35: number analyzed (Participants) | 29 | 35
  Calcium; Post-infusion assessment, n=29, 35 | 0.018 (0.0953) | 0.023 (0.0861)
  Calcium; early withdrawal, n=1, 1: number analyzed (Participants) | 1 | 1
  Calcium; early withdrawal, n=1, 1 | -0.120 (NA) — NA indicates standard deviation was not calculable for a single data point. | -0.230 (NA) — NA indicates standard deviation was not calculable for a single data point.
  Chloride; Day 2, n=35, 35: number analyzed (Participants) | 35 | 35
  Chloride; Day 2, n=35, 35 | 1.5 (2.02) | 1.4 (2.03)
  Chloride; Post-infusion assessment, n=30, 35: number analyzed (Participants) | 30 | 35
  Chloride; Post-infusion assessment, n=30, 35 | -1.5 (1.83) | -1.3 (2.63)
  Chloride; early withdrawal, n=1, 1: number analyzed (Participants) | 1 | 1
  Chloride; early withdrawal, n=1, 1 | 2.0 (NA) — NA indicates standard deviation was not calculable for a single data point. | 8.0 (NA) — NA indicates standard deviation was not calculable for a single data point.
  Carbon dioxide; Day 2, n=34, 35: number analyzed (Participants) | 34 | 35
  Carbon dioxide; Day 2, n=34, 35 | 0.7 (2.34) | 0.3 (2.63)
  Carbon dioxide, Post-infusion assessment, n=29,35: number analyzed (Participants) | 29 | 35
  Carbon dioxide, Post-infusion assessment, n=29,35 | 1.9 (2.06) | 1.9 (2.67)
  Carbon dioxide, early withdrawal, n=1, 1: number analyzed (Participants) | 1 | 1
  Carbon dioxide, early withdrawal, n=1, 1 | -2.0 (NA) — NA indicates standard deviation was not calculable for a single data point. | 6.0 (NA) — NA indicates standard deviation was not calculable for a single data point.
  Glucose; Day 2, n=35,35: number analyzed (Participants) | 35 | 35
  Glucose; Day 2, n=35,35 | 0.13 (2.013) | 1.51 (2.156)
  Glucose; Post-infusion assessment, n=30, 35: number analyzed (Participants) | 30 | 35
  Glucose; Post-infusion assessment, n=30, 35 | -0.70 (1.994) | -0.35 (2.283)
  Glucose; early withdrawal, n= 1, 1: number analyzed (Participants) | 1 | 1
  Glucose; early withdrawal, n= 1, 1 | 0.70 (NA) — NA indicates standard deviation was not calculable for a single data point. | -5.20 (NA) — NA indicates standard deviation was not calculable for a single data point.
  Potassium; Day 2, n= 34, 35: number analyzed (Participants) | 34 | 35
  Potassium; Day 2, n= 34, 35 | 0.06 (0.392) | -0.06 (0.346)
  Potassium; Post-infusion assessment, n= 29, 35: number analyzed (Participants) | 29 | 35
  Potassium; Post-infusion assessment, n= 29, 35 | 0.21 (0.362) | 0.18 (0.355)
  Potassium; early withdrawal, n= 1,1: number analyzed (Participants) | 1 | 1
  Potassium; early withdrawal, n= 1,1 | -0.10 (NA) — NA indicates standard deviation was not calculable for a single data point. | 0.50 (NA) — NA indicates standard deviation was not calculable for a single data point.
  Magnesium; Day 2, n= 35,35: number analyzed (Participants) | 35 | 35
  Magnesium; Day 2, n= 35,35 | 0.073 (0.2098) | -0.003 (0.0657)
  Magnesium, Post-infusion assessment, n= 30,35: number analyzed (Participants) | 30 | 35
  Magnesium, Post-infusion assessment, n= 30,35 | 0.026 (0.0760) | 0.009 (0.0772)
  Magnesium; early withdrawal, n= 1,1: number analyzed (Participants) | 1 | 1
  Magnesium; early withdrawal, n= 1,1 | -0.060 (NA) — NA indicates standard deviation was not calculable for a single data point. | 0.030 (NA) — NA indicates standard deviation was not calculable for a single data point.
  Phosphate; Day 2, n= 35,35: number analyzed (Participants) | 35 | 35
  Phosphate; Day 2, n= 35,35 | -0.101 (0.2684) | -0.170 (0.2357)
  Phosphate; Post-infusion assessment, n= 30,35: number analyzed (Participants) | 30 | 35
  Phosphate; Post-infusion assessment, n= 30,35 | 0.041 (0.2267) | 0.094 (0.2864)
  Phosphate; early withdrawal, n= 1,1: number analyzed (Participants) | 1 | 1
  Phosphate; early withdrawal, n= 1,1 | 0.100 (NA) — NA indicates standard deviation was not calculable for a single data point. | -0.120 (NA) — NA indicates standard deviation was not calculable for a single data point.
  Sodium; Day 2, n= 35,35: number analyzed (Participants) | 35 | 35
  Sodium; Day 2, n= 35,35 | 0.7 (2.13) | 0.1 (1.69)
  Sodium; Post-infusion assessment, n= 30,35: number analyzed (Participants) | 30 | 35
  Sodium; Post-infusion assessment, n= 30,35 | -1.1 (2.05) | -0.2 (2.11)
  Sodium; early withdrawal, n= 1,1: number analyzed (Participants) | 1 | 1
  Sodium; early withdrawal, n= 1,1 | -1.0 (NA) — NA indicates standard deviation was not calculable for a single data point. | 3.0 (NA) — NA indicates standard deviation was not calculable for a single data point.

28. Secondary Outcome: Change From Baseline in Direct Bilirubin, Bilirubin, Indirect Bilirubin, Creatinine and Urate Levels in Maternal Participants
Description: Blood samples were collected for the evaluation of change from Baseline in levels of direct bilirubin, bilirubin, indirect bilirubin, creatinine and urate. Baseline is defined as the last available assessment prior to the first dose of study treatment. Change from Baseline is the post-dose visit value minus Baseline. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title). NA indicates standard deviation was not calculable for a single data point.
Time Frame: Baseline and up to 1 week
Population: Maternal Safety Population
Measure: Mean (Standard Deviation); unit: micromoles per liter (µmol/L)
Arm/Group | Retosiban | Atosiban
Number analyzed (Participants) | 47 | 50
micromoles per liter (µmol/L)
  Direct Bilirubin; Day2, n=35,35: number analyzed (Participants) | 35 | 35
  Direct Bilirubin; Day2, n=35,35 | -0.3 (0.85) | -0.3 (0.66)
  Post-infusion assessment, n=30,35: number analyzed (Participants) | 30 | 35
  Post-infusion assessment, n=30,35 | -0.5 (3.41) | -0.1 (0.73)
  Direct Bilirubin;early withdrawal, n=1,1: number analyzed (Participants) | 1 | 1
  Direct Bilirubin;early withdrawal, n=1,1 | 0.0 (NA) — NA indicates standard deviation was not calculable for a single data point. | 0.0 (NA) — NA indicates standard deviation was not calculable for a single data point.
  Bilirubin;Day2, n= 35,35: number analyzed (Participants) | 35 | 35
  Bilirubin;Day2, n= 35,35 | -0.7 (2.52) | -1.3 (2.03)
  Bilirubin; Post-infusion assessment, n= 30, 35: number analyzed (Participants) | 30 | 35
  Bilirubin; Post-infusion assessment, n= 30, 35 | -1.1 (8.24) | -0.5 (2.01)
  Bilirubin; early withdrawal, n= 1,1: number analyzed (Participants) | 1 | 1
  Bilirubin; early withdrawal, n= 1,1 | -2.0 (NA) — NA indicates standard deviation was not calculable for a single data point. | -3.0 (NA) — NA indicates standard deviation was not calculable for a single data point.
  Indirect Bilirubin; Day2, n=35,35: number analyzed (Participants) | 35 | 35
  Indirect Bilirubin; Day2, n=35,35 | -0.4 (2.35) | -1.1 (1.98)
  Indirect Bilirubin;Postinfusion assessment,n=30,35: number analyzed (Participants) | 30 | 35
  Indirect Bilirubin;Postinfusion assessment,n=30,35 | -0.6 (5.06) | -0.4 (2.03)
  Indirect Bilirubin; early withdrawal, n=1,1: number analyzed (Participants) | 1 | 1
  Indirect Bilirubin; early withdrawal, n=1,1 | -2.0 (NA) — NA indicates standard deviation was not calculable for a single data point. | -3.0 (NA) — NA indicates standard deviation was not calculable for a single data point.
  Creatinine; Day2, n=35,34: number analyzed (Participants) | 35 | 34
  Creatinine; Day2, n=35,34 | 1.75 (6.765) | 0.04 (5.336)
  Creatinine; Post-infusion assessment, n=30,33: number analyzed (Participants) | 30 | 33
  Creatinine; Post-infusion assessment, n=30,33 | 2.19 (4.437) | 0.72 (4.680)
  Creatinine; early withdrawal, n=1,1: number analyzed (Participants) | 1 | 1
  Creatinine; early withdrawal, n=1,1 | -0.90 (NA) — NA indicates standard deviation was not calculable for a single data point. | -6.10 (NA) — NA indicates standard deviation was not calculable for a single data point.

29. Secondary Outcome: Number of Maternal Participants With AEs of Special Interest (AESI)
Description: Maternal AESI included: maternal death; chorioamnionitis and its complications (clinical chorioamnionitis, preterm premature rupture of membranes, endomyometritis, wound infection, pelvic abscess, bacteremia, septic shock, disseminated intravascular coagulation, and adult RDS); placental abruption; postpartum hemorrhage - postpartum hemorrhage and/or retained placenta and pulmonary edema. The number of participants with at least one AESI has been presented.
Time Frame: Up to 6 weeks post-delivery
Population: Maternal Safety Population
Measure: Number; unit: Participants
Arm/Group | Retosiban | Atosiban
Number analyzed (Participants) | 47 | 50
Participants | 4 | 7

30. Secondary Outcome: Number of Maternal Participants With Disease Related AEs (DRE)
Description: Maternal DREs included: signs and symptoms of labor discomfort (example, cramping, backache, muscle aches, nausea); subsequent episodes of preterm labor and hospitalization for delivery. The number of participants with at least one DRE has been presented.
Time Frame: Up to 6 weeks post-delivery
Population: Maternal Safety Population
Measure: Number; unit: Participants
Arm/Group | Retosiban | Atosiban
Number analyzed (Participants) | 47 | 50
Participants | 5 | 5

31. Secondary Outcome: Number of Participants With Fetal Non-serious AEs and SAEs
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose: results in death; is life threatening; requires hospitalization or prolongation of existing hospitalization; results in disability/incapacity; is a congenital anomaly/birth defect; important medical events that may require medical or surgical intervention to prevent one of the other outcomes described before; is associated with liver injury and impaired liver function. The number of participants who experienced at least one non-serious AE and one SAE has been presented.
Time Frame: Up to 17 weeks
Population: Maternal Safety Population
Measure: Number; unit: Participants
Arm/Group | Retosiban | Atosiban
Number analyzed (Participants) | 47 | 50
Participants
  Non-serious AE | 6 | 6
  SAE | 4 | 2

32. Secondary Outcome: Number of Participants With Fetal AESI
Description: Fetal AESI included: intrauterine fetal demise; category II or III fetal heart rate tracing; and fetal inflammatory response syndrome characterized by cord blood interleukin-6 >11 picogram per milliliter (pg/mL), funisitis, or chorionic vasculitis. The number of participants who experienced at least one AESI has been presented.
Time Frame: Up to 17 weeks
Population: Maternal Safety Population
Measure: Number; unit: Participants
Arm/Group | Retosiban | Atosiban
Number analyzed (Participants) | 47 | 50
Participants | 5 | 5

33. Secondary Outcome: Neonatal APGAR Scores
Description: APGAR is a quick test to assess the health of new born children. The test is performed at 1 and 5 minutes after birth. APGAR scale is determined by evaluating the new born on five categories (appearance, pulse, grimace, activity and respiration) on a scale from zero to two, then summing up the five values obtained. APGAR score ranges from 0 to 10 where a score of 7 and above is normal. The mean and standard deviation of APGAR scores at one minute and at five minutes of birth has been presented.Only those participants with data available at the specified data points were analyzed.
Time Frame: Up to 5 minutes after birth
Population: Neonatal ITT Population
Measure: Mean (Standard Deviation); unit: Score on APGAR scale
Arm/Group | Retosiban | Atosiban
Number analyzed (Participants) | 47 | 50
Score on APGAR scale
  one minute, n=46, 50: number analyzed (Participants) | 46 | 50
  one minute, n=46, 50 | 8.2 (1.35) | 8.4 (1.14)
  five minutes, n=46, 50: number analyzed (Participants) | 46 | 50
  five minutes, n=46, 50 | 9.1 (0.96) | 9.4 (0.67)

34. Secondary Outcome: Weight of Neonates
Description: The weight of neonates was obtained from the neonate birth record. The mean weight of neonates and standard deviation has been presented. Only those participants with data available at the specified data points were analyzed.
Time Frame: Up to 17 weeks
Population: Neonatal ITT Population
Measure: Mean (Standard Deviation); unit: grams (g)
Arm/Group | Retosiban | Atosiban
Number analyzed (Participants) | 46 | 49
grams (g) | 2761.9 (567.84) | 2844.4 (664.80)

35. Secondary Outcome: Head Circumference of Neonates
Description: The head circumference was determined from the neonate birth record. Only those participants with data available at the specified data points were analyzed.
Time Frame: Up to 17 weeks
Population: Neonatal ITT Population
Measure: Mean (Standard Deviation); unit: centimeters (cm)
Arm/Group | Retosiban | Atosiban
Number analyzed (Participants) | 43 | 42
centimeters (cm) | 32.95 (2.179) | 33.00 (1.892)

36. Secondary Outcome: Number of Neonatal Participants With Non-serious AEs and SAEs
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose: results in death; is life threatening; requires hospitalization or prolongation of existing hospitalization; results in disability/incapacity; is a congenital anomaly/birth defect; important medical events that may require medical or surgical intervention to prevent one of the other outcomes described before; is associated with liver injury and impaired liver function. The number of participants who experienced at least one non-serious AE and one SAE has been presented. Neonatal Safety Population consisted of neonates whose mothers received randomized treatment.
Time Frame: Up to 28 days after the EDD of 40 weeks gestation
Population: Neonatal Safety Population
Measure: Number; unit: Participants
Arm/Group | Retosiban | Atosiban
Number analyzed (Participants) | 47 | 50
Participants
  Non-serious AEs | 23 | 17
  SAEs | 10 | 11

37. Secondary Outcome: Number of Neonatal Participants With AESI
Description: Neonatal AESI included: Neonatal death; Asphyxia; Infections (early onset neonatal sepsis, septic shock, pneumonia, meningitis); RDS; Hypotension; IVH/periventricular leukomalacia; Bronchopulmonary dysplasia; Neonatal acidosis; Hyperbilirubinemia; Necrotizing enterocolitis; and Hypoxic ischemic encephalopathy. The number of neonatal participants who experienced at least one AESI has been presented.
Time Frame: Up to 28 days after EDD of 40 weeks gestation
Population: Neonatal Safety Population
Measure: Number; unit: Participants
Arm/Group | Retosiban | Atosiban
Number analyzed (Participants) | 47 | 50
Participants | 19 | 16

38. Secondary Outcome: Number of Neonatal Participants With DRE
Description: The disease related neonatal events occurring in Infants born prior to 37 completed weeks included: apnea (severe), respiratory failure due to fatigue, hypoxia, or air leak from alveolar injury, patent ductus arteriosus, bradycardia, ventriculomegaly, cerebellar hemorrhage, hydrocephalus other than congenital, gastroesophageal reflux, aspiration pneumonia, anemia, retinopathy of prematurity (all stages), hearing disorder, temperature instability and hypoglycemia. The number of participants with at least one DRE has been presented.
Time Frame: Up to 28 days after EDD of 40 weeks gestation
Population: Neonatal Safety Population
Measure: Number; unit: Participants
Arm/Group | Retosiban | Atosiban
Number analyzed (Participants) | 47 | 50
Participants | 5 | 3

39. Secondary Outcome: Maternal Length of Stay in Hospital
Description: The length of hospital stay associated with hospital admission for preterm labor and term labor/term delivery was collected from review of medical records. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title).
Time Frame: Up to 28 days post EDD (40 0/7 weeks gestation)
Population: Maternal Safety Population
Measure: Median (Full Range); unit: Days
Arm/Group | Retosiban | Atosiban
Number analyzed (Participants) | 47 | 50
Days
  Preterm labor, n=13, 10: number analyzed (Participants) | 13 | 10
  Preterm labor, n=13, 10 | 5.549 [1.32 to 72.00] | 7.487 [0.87 to 37.82]
  Term labor, n=25, 28: number analyzed (Participants) | 25 | 28
  Term labor, n=25, 28 | 3.146 [0.17 to 62.71] | 3.398 [0.41 to 36.74]

40. Secondary Outcome: Number of Participants Admitted to Particular Hospital Unit
Description: Maternal healthcare resource utilization associated with an episode of preterm labor and normal term delivery were collected from the review of medical records. The number of participants who were admitted to a particular hospital unit like general ward, private/semi-private room, recovery, and other has been presented.
Time Frame: Up to 28 days post EDD (40 0/7 weeks gestation)
Population: Maternal Safety Population
Measure: Number; unit: Participants
Arm/Group | Retosiban | Atosiban
Number analyzed (Participants) | 47 | 50
Participants
  Preterm labor, general ward | 9 | 7
  Preterm labor, private/semi-private room | 1 | 0
  Preterm, Other | 3 | 4
  Normal term labor, general ward | 16 | 12
  Normal term labor, ward-not specified | 2 | 0
  Normal term labor,private/semi-private room | 1 | 7
  Normal term labor, recovery | 1 | 2
  Normal term labor, Other | 5 | 7

41. Secondary Outcome: Retosiban Clearance
Description: Maternal blood samples were collected at the indicated time points for pharmacokinetic analysis. Data is a combined data set. Data is presented for 10 participants from retosiban arm of study 200719 (NCT02377466) and 43 participants from retosiban arm of study 200721 (NCT02292771).
Time Frame: Day 1 (2 to 4 hours, 10 to 14 hours) and Day 2 (22 to 26 hours, and 48 to 54 hours) post-infusion
Population: Maternal Safety Population. Data is a combined data set. Data is presented for 10 participants from retosiban arm of study 200719 (NCT02377466) and 43 participants from retosiban arm of study 200721 (NCT02292771).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour
Arm/Group | Retosiban
Number analyzed (Participants) | 53
Liters per hour | 83.4 (5.25)

42. Secondary Outcome: Volume of Distribution of Retosiban
Description: as for outcome 41
Time Frame: Day 1 (2 to 4 hours, 10 to 14 hours) and Day 2 (22 to 26 hours, and 48 to 54 hours) post-infusion
Population: as for outcome 41
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Retosiban
Number analyzed (Participants) | 53
Liters | 68.6 (109)

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from the start of study treatment and until Day 894.
Description: SAEs and AEs were analyzed in Maternal Safety Population and Neonatal Safety Population which comprised of mothers randomly assigned to treatment who were exposed to study treatment and neonates whose mothers received randomized treatment. One participant was withdrawn prior to delivery and was not included in the summary.
Groups:
- Retosiban (Maternal); Retosiban (Fetal); Retosiban (Neonatal): Participants were administered 6 milligram (mg) IV loading dose of retosiban over 5 minutes followed by a 6 milligram per hour (mg/hour) continuous infusion of retosiban over 48 hours. Participants with an inadequate response any time after first hour of treatment were administered another 6 mg retosiban loading dose followed by 12 mg/hour continuous infusion for remainder of 48-hour treatment period.
- Atosiban (Maternal); Atosiban (Fetal); Atosiban (Neonatal): Participants were administered atosiban in 3 successive stages. An initial bolus dose of 6.75 mg using atosiban 6.75 mg/0.9 milliliter (mL) solution for injection, followed by continuous high dose infusion at 18 mg/hour for 3 hours, then a lower 6 mg/hour infusion for the remainder of the 48-hour using the atosiban 37.5 mg/5 mL concentrate for solution.
Arm/Group | Retosiban (Maternal) | Atosiban (Maternal) | Retosiban (Fetal) | Atosiban (Fetal) | Retosiban (Neonatal) | Atosiban (Neonatal)
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/50 | 0/47 | 0/50 | 0/46 | 1/50
Serious Adverse Events (participants affected / at risk) | 7/47 | 9/50 | 4/47 | 2/50 | 10/46 | 11/50
Other Adverse Events (participants affected / at risk) | 34/47 | 25/50 | 6/47 | 6/50 | 23/46 | 17/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Retosiban (Maternal) (N=47) | Atosiban (Maternal) (N=50) | Retosiban (Fetal) (N=47) | Atosiban (Fetal) (N=50) | Retosiban (Neonatal) (N=46) | Atosiban (Neonatal) (N=50)
Postpartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Preterm premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Normal labour (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Premature labour (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Premature separation of placenta (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oligohydramnios (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hydrops foetalis (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Amniotic cavity infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial disease carrier (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia neonatal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 3 (3)
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foetal monitoring abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Foetal heart rate disorder (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Foetal heart rate deceleration abnormality (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Congenital hydronephrosis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ankyloglossia congenital (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial septal defect (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cataract congenital (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyloric stenosis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ventricular septal defect (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neonatal respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Choking (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Meconium aspiration syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sudden infant death syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Milk allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Retosiban (Maternal) (N=47) | Atosiban (Maternal) (N=50) | Retosiban (Fetal) (N=47) | Atosiban (Fetal) (N=50) | Retosiban (Neonatal) (N=46) | Atosiban (Neonatal) (N=50)
Foetal heart rate disorder (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Foetal heart rate deceleration abnormality (Cardiac disorders) | 0 (0) | 0 (0) | 3 (15) | 0 (0) | 0 (0) | 0 (0)
Bradycardia foetal (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia foetal (Cardiac disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Foetal hypokinesia (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Oligohydramnios (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Postpartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Polyhydramnios (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Premature labour (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Preterm premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Cephalhaematoma (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperbilirubinaemia neonatal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 10 (10) | 8 (8)
Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neonatal respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient tachypnoea of the newborn (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Choking (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory disorder neonatal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Use of accessory respiratory muscles (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infantile colic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 10 (12) | 5 (5) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Regurgitation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal rigidity (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 4 (4) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial vaginosis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervicitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asymptomatic bacteriuria (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginitis gardnerella (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Genital candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulpitis dental (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyuria (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Skin candida (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ureaplasma infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scrotal oedema (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Testicular retraction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 (4) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast engorgement (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine atony (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulval oedema (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Polycythaemia neonatorum (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia of pregnancy (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Auditory disorder (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eyelid oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Generalised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suprapubic pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelid haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 8 (8) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Burning sensation (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia test positive (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psychiatric evaluation abnormal (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Candida test positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Klebsiella test positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mood swings (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acne infantile (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Macule (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Congenital hydronephrosis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hydrocele (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal pain (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-10-04): https://cdn.clinicaltrials.gov/large-docs/71/NCT02292771/SAP_000.pdf
  • Study Protocol (2016-12-21): https://cdn.clinicaltrials.gov/large-docs/71/NCT02292771/Prot_001.pdf